CLINICAL TRIAL: NCT03153280
Title: A Phase Ib, Dose Escalation Study of Lithium When Added to Standard Chemotherapy of Oxaliplatin and Capecitabine in Patients With Advanced Oesophago-Gastric or Colorectal Cancer
Brief Title: Dose Escalation Study of Lithium With Oxaliplatin and Capecitabine in Advanced Oesophago-Gastric or Colorectal Cancer
Acronym: Lithium
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Poor accrual and the field has moved on.
Sponsor: Cancer Trials Ireland (Network)
Collaborators: University College Cork (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTRIAL-IE (ICORG) 11-32; 2014-000186-47 (EudraCT Number)
Record Dates: First submitted 2017-05-10; First posted 2017-05-15 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Neoplasms; Stomach Neoplasm; Esophageal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms; Stomach Neoplasms; Esophageal Neoplasms | interventions — Lithium; Oxaliplatin; Capecitabine

STUDY DESIGN:
Intervention Model Description: Lithium: starting dose: 2x 400mg p.o. per day. Initial target blood concentration (Level 1 = 0.6mmol/L).
  Oxaliplatin: 130 mg/m2 in 500 ml normal saline (NS) over 120 minutes on Day 1 of each 3 week cycle.
  Capecitabine: 1000 mg/m2 b.i.d po on Days 1 to 14 of each 3 week cycle.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lithium, Oxaliplatin & Capecitabine (Experimental): Target serum concentrations of escalating doses of lithium (0.6, 0.9, 1.26 or 1.4 mmol/L) in combination standard chemotherapy - oxaliplatin and capecitabine.
  Interventions: Drug: Lithium; Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: Lithium — Dose escalation of Lithium to determine the maximum tolerated dose (MTD)
Drug: Oxaliplatin — Dose as used in standard of care - 130 mg/m2.
Drug: Capecitabine — Dose as used in standard of care - 800 - 1000 mg/m2

SUMMARY:
This study is a phase Ib, open label, multi-centre trial designed to estimate the Maximum Tolerated Dose (MTD) of lithium when combined with a standard chemotherapy regimen of oxaliplatin and capecitabine in patients with advanced, unresectable, oesophago-gastric or colorectal cancer who have received no previous treatment for advanced disease (previous adjuvant or neo-adjuvant treatment is acceptable if completed at least 6 months prior to registration).

The study follows a modified Fibonacci, 3+3, dose escalation design. Patients are enrolled in cohorts of 3. All three patients in each cohort must complete at least two cycles of treatment to be evaluable for toxicity. If a patient cannot complete 2 cycles, another patient will be enrolled.

DETAILED DESCRIPTION:
This study is a Phase Ib, open label, multi-centre, dose escalation trial to assess the dose of lithium that can be safely combined with standard treatment oxaliplatin and capecitabine chemotherapy.

Registered patients will be treated with lithium combined with a standard chemotherapy regimen of oxaliplatin and capecitabine until a maximum of 6 x 21 day cycles (18 weeks), tumour progression, unacceptable toxicity, pregnancy, withdrawal of consent or withdrawal at the discretion of the investigator, whichever occurs first.

After discontinuation of study treatment, all patients will be followed for safety for at least 30 days.

Patients who discontinue treatment for reasons other than disease progression will continue to be followed every 9 weeks in accordance with standard of care for efficacy (i.e. tumour assessment) until disease progression, death, withdrawal of consent, loss to follow up or until the start of a new anti-neoplastic treatment, whichever occurs first.

Once the patient has documented disease progression, they will be followed up every three months (±1 month) for survival status.

The trial will be a traditional 3+3 design: cohorts of 3 patients will be treated with lithium combined with standard treatment oxaliplatin and capecitabine chemotherapy.

The doses of oxaliplatin and capecitabine have been established in prior phase II and III studies and will not be escalated. Lithium target serum concentrations are assigned at registration according to a defined dose escalation scheme. Study lithium dose escalation will follow a modified Fibonacci 3+3 sequence.

A -1 dose level (0.4mmol/L) is included in case dose de-escalation is needed.

The levels of lithium achieved in each patient will be established by regular assessment of steady state serum concentrations.

Lithium will start at a low level and dose escalations will be performed in cohorts of 3 patients according to a standard 3+3 algorithm.

Dose escalation and determination of MTD will be based on the occurrence of Dose Limiting Toxicities (DLT) as defined below.

The first cohort of 3 patients will commence at dose level 1. All patients in each cohort will be observed for two cycles on the specified dose:

* If none of 3 patients at a given dose level experiences a DLT, accrual will continue to the next dose level according to the protocol.
* If 1 of 3 patients experiences a DLT at a given dose level, 3 additional patients will be treated at the same dose. If no additional patient has a DLT in this cohort, accrual will continue to the next dose level according to the protocol.
* If 2 or more patients in 3 or 6 patients treated at a given dose experience a DLT, the next lowest dose level will define the MTD.

A Dose Limiting Toxicity (DLT) is defined as any of the following adverse events occurring during the two first cycles (within 42 days from first dose) of treatment and possibly, probably or definitely related to the combination of lithium, oxaliplatin and capecitabine:

A. Grade 3 or 4 non-haematological toxicity other than nausea, vomiting or fatigue.

B. Grade 3 or 4 thrombocytopenia: grade 4 thrombocytopenia (platelet count < 25 x 109/L) or grade 3/4 thrombocytopenia (grade 3 platelet count: 25 x 109/L to < 50 x 109/L) associated with bleeding.

C. Complicated grade 4 neutropenia (< 0.5 x 109/L): fever, sepsis > 5 days of duration.

D. Any significant* grade 2 and higher toxicity other than nausea, vomiting, rash, alopecia or anaemia that persists longer than 35 days after the start of cycle 1.

*"Significant" defined as affecting quality of life or patient safety as determined by investigator.

Clinical and laboratory parameters will be assessed to evaluate disease response and toxicity of study therapy. Safety assessments will be performed every 3 weeks for the 18 weeks. Efficacy assessments (Radiological examination) will be performed on all patients every 9 weeks (+/- 1 week).

An End of Treatment visit will be performed for patients within 30 days (+/- 1 week) post last dose or disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be given according to ICH/GCP and national/local regulations, and be obtained prior to any study-related procedures.
2. Histologically or cytologically confirmed adenocarcinoma of the colon, rectum, stomach, gastro-oesophageal junction or lower third of the oesophagus.
3. Metastatic disease not amenable to surgical resection with curative intent.
4. Eastern Co-operative Oncology Group (ECOG) performance status 2 (Appendix B).
5. Age ≥ to 18.
6. Estimated life expectancy ≥ 3 months.
7. Measurable disease, defined as at least 1 uni-dimensionally measurable lesion on a CT scan as defined by RECIST criteria, Version 1.1 (Appendix F).
8. Adequate haematological, hepatic, and renal function defined as:

   a. Renal: i. Calculated creatinine clearance (CrCl) 50ml/min (see Appendix G) b. Liver function tests: i. Total Bilirubin ≤ ULN ii. ALT and AST ≤ 2.5 x ULN (≤ 5 x ULN with liver involvement of their cancer) iii. Alkaline Phosphatase ≤ 2.5 x ULN (≤ 5 x ULN with liver involvement of their cancer) c. Haematology: i. Haemoglobin 9.0 g/dL for females and 10.0 g/dL for males ii. Absolute neutrophil count 1.5 x 109/L iii. Platelet count 100 x109/L
9. Normal thyroid function (TSH 0.4-3.5mUL).
10. Able to swallow and retain oral medication.
11. Women of child-bearing potential and male patients must agree to use adequate contraception for the duration of study participation and for up to 3 months following discontinuation of therapy. Adequate contraception is defined as any medically recommended (or combination of methods) as per standard of care.
12. Women of child bearing potential must have pregnancy excluded by urine or serum beta-HCG testing within 7 days prior to registration.

Exclusion Criteria:

1. Received prior chemotherapy for metastatic disease. (Patients who received prior adjuvant or neo-adjuvant chemotherapy or definitive radio-chemotherapy for localised disease are eligible if the chemotherapy has stopped at least 6 months before registration).
2. Previous or concurrent malignancy within the past 5 years, with the exception of basal cell carcinoma of the skin or in-situ neoplasia of the uterine cervix or bladder.
3. Brain or other Central Nervous System (CNS) metastases.
4. Known di-hydropyrimidine dehydrogenase (DPD) deficiency.
5. Screening electrocardiogram (ECG) with evidence of:

   1. QT prolongation (QTc > 450 ms in males and > 470 ms in females)
   2. 2nd or 3rd degree heart block
   3. Other severe cardiac dysfunction (ECG must be assessed for all patients within 14 days prior to registration)
6. Clinically significant cardiovascular disease including:

   1. Cerebrovascular accident within 6 months prior to registration
   2. Myocardial infarction within 6 months prior to registration
   3. Uncontrolled angina
   4. Uncontrolled hypertension
   5. Clinically significant valvular disease
   6. Congestive Heart Failure (NYHA Class 2) (See Appendix E).
7. Severe chronic obstructive pulmonary disease (COPD) > Grade 2 according to NCI CTCAE v4.0.
8. Known history or family history of Brugada Syndrome.
9. Symptoms or signs of peripheral neuropathy.
10. Ongoing infection > Grade 2 according to NCI CTCAE v4.0.
11. Seizure disorder requiring medication.
12. Dehydration Grade 1 according to NCI CTCAE v4.0; patients on Low sodium diet; Addison's disease.
13. Known hypersensitivity to lithium, oxaliplatin or fluoropyrimidines.
14. Pregnant or nursing women.
15. Concurrent treatment with any other investigational agents within 30 days prior to registration.
16. Any psychological, physical, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; (those conditions should be discussed with the patient before registration in the trial).
17. Unable or unwilling to discontinue (and substitute if necessary) use of prohibited medications for at least 30 days prior to and for the duration of study treatment (see section 7.5 for a description of prohibited medications).
18. Patients weighing less than 50kg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-01-13 (Actual); Primary Completion 2023-09-07 (Actual); Study Completion 2023-09-07 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLT) within the two first cycles at each dose level. | 26 months
  The MTD will be based on the incidence of DLT within the two first cycles of lithium in combination with standard chemotherapy of oxaliplatin and capecitabine at each dose level.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) as defined by RECIST Criteria Version 1.1. | 3 years
  PFS will be defined as the time from the start of treatment until disease progression or death as a result of any cause.
Objective Response Rate (ORR) as defined by RECIST Criteria Version 1.1. | 3 years
  ORR is defined as the proportion of patients who receive a Complete Response or a Partial Response (CR + PR).
Incidence of adverse events reported as per the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0. (Safety and Tolerability). | 3 years
  Safety will be assessed by standard clinical and laboratory tests.

CONTACTS AND LOCATIONS:
Overall Officials: Cancer Trials Ireland Dublin 11, Ireland, Study Director — Cancer Trials Ireland
Locations (2):
- Ireland (2):
  - Cork University Hospital, Cork
  - St James's Hospital, Dublin

IPD SHARING:
Plan to Share IPD: No